CLINICAL TRIAL: NCT06627439
Title: Comadres Saludables: A Web-Based Promotora Training Program for Obesity Prevention in Hispanic Women
Brief Title: A Web-Based Healthy Living Training for Promotores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISA Associates, Inc. (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44MD016228 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity Prevention
Keywords: Obesity; Latina
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based Comadres Saludables CHW Training (Experimental): Experimental group participants will have access to the web-based Comadres Saludables training for three months.
  Interventions: Behavioral: Comadres Saludables
- HHS Promoting Healthy Choices and Community Changes (Active Comparator): Control condition participants will receive information on how to access the HHS CHW Promoting Healthy Choices and Community Changes training. They will be asked to review for three months.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Comadres Saludables — Comadres Saludables is a web-based healthy living training for community health workers aimed at addressing obesity in Latinas. Comadres Saludables will combine both theory and evidence-based practices to provide participants with the self-efficacy, knowledge, and skills required to effectively implement an obesity intervention for Hispanic women. Participants (CHWs) will build their skillset through interactive quizzes, exercises, and video role-playing scenarios. Additionally, Comadres Saludables allows participants to utilize interactive mHealth tools to enhance implementation with Hispanic women. Participants will access the training for three months.
  Arms: Web-based Comadres Saludables CHW Training
Behavioral: Control — Participants will access the web-based HHS Promoting Healthy Choices and Community Changes that includes a variety of content via text, audio, and video. The information is designed to educate CHWs on how to implement health interventions for positive community change. They are asked to review it for three months.
  Arms: HHS Promoting Healthy Choices and Community Changes

SUMMARY:
The goal of this clinical trial is to test a new web-based promotora de salud/ community health worker (CHW) training. This training is designed to provide CHWs with the knowledge and skills to effectively implement a healthy living intervention for Latinas. The main question it aims to answer is:

o Do CHWs who complete the web-based healthy living training have higher self-efficacy in implementing core lifestyle intervention learning components for obesity interventions in Hispanics than CHWs who do not?

Participants will:

* Complete a baseline survey asking about self-efficacy related to implementing core lifestyle intervention learning components, knowledge, health behaviors, and skill mastery.
* Be randomized to receive the new web-based training or to a standard CHW training designed by Health and Human Services. The new web-based training provides promotores with the self-efficacy, knowledge, and skills required to effectively implement an obesity intervention for Hispanic women. Promotores will build their skillset through interactive quizzes, exercises, video role-playing scenarios, and interactive tools.
* Complete follow-up surveys at 3 months and 6 months after the baseline survey. This survey will ask the same questions as the baseline survey and will include additional questions regarding satisfaction with training and behavior application.

Researchers will compare participants who receive the new web-based training to participants who utilize the HHS training. The goal is to see whether the new web-based training increases self-efficacy among CHWs to effectively implement core lifestyle learning components for obesity interventions in Hispanics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and old
* Comfortable speaking, reading, and writing English OR Spanish
* Female
* Access to a computer that has internet
* Not Pregnant
* Have a community health worker certification through the state of TX OR have worked over 6 moths as a community health worker and meets core competencies for CHWs
* Provides services to Hispanic populations

Exclusion Criteria:

* Less than 18 years of age and old
* Not comfortable speaking, reading, and writing English OR Spanish
* Male
* Does not have access to a computer that has internet
* Pregnant
* Does not have a community health worker certification through the state of TX OR have not worked over 6 moths as a community health worker and does not meet core competencies for CHWs
* Does not provide services to Hispanic populations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Self-Efficacy at week 12 and week 24 | Baseline, Week 12, and Week 24
  19-item questionnaire that measures the degree to which an individual perceives self efficacy in implementing core lifestyle intervention learning components for obesity interventions in Hispanics. Score ranges from 19-133 with a higher score indicating higher self-efficacy.

SECONDARY OUTCOMES:
Obesity Intervention Knowledge Questionnaire | Baseline, Week 12, and Week 24
  Measured using 40 questions developed specifically for the proposed study. Items measure knowledge acquired about the healthy living intervention and are averaged to form a score ranging from 1 to 40, where higher scores indicate higher knowledge.
Self-Report Skill Mastery | Baseline, Week 12, and Week 24
  Measured using 15-items that assess self-report skill mastery across three scenarios. Participants rate their skill mastery on a scale of 1 (strongly disagree) to 5 (strongly agree) they have the skills to performs specific tasks. Score ranges from 5 to 75 with higher scores indicating higher self-report skill mastery.
Satisfaction with Training | Week 12
  Measured using 21-items that assess an individuals satisfaction with using the web-based CHW training. Score ranges from 21 to 105 with higher scores indicating higher satisfaction.
Behavior Application | Week 24
  Measured using 20-items that assess whether an individual has utilized the knowledge and skills learned in the training in their day-to-day work life. Score ranges from 20 to 100 with higher scores indicating higher usage of the knowledge and skills.

CONTACTS AND LOCATIONS:
Overall Officials: Debra M Rios, DrPH, Principal Investigator — ISA Associates
Locations (1):
- ISA Associates, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No